CLINICAL TRIAL: NCT01635543
Title: Investigation of Sexual Function in Crohn's Disease Patients With Perianal Fistulas
Status: Withdrawn | Type: Observational
Why Stopped: This study was terminated due to some challenges in recruitment process
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H11-01890
Record Dates: First submitted 2012-06-27; First posted 2012-07-09 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-10

CONDITIONS: Crohn's Disease; Peri-anal Fistulas; Sexual Dysfunction
MeSH Terms: conditions — Crohn Disease; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Crohn's Disease with peri-anal fistulas: Identifying Crohn's Disease patients with peri-anal fistulas and suffering from sexual dysfunction.

SUMMARY:
Objective:

The aim of this study is to investigate whether Crohn's Disease patients with peri-anal fistulas will suffer from sexual dysfunction in an attempt to help us identify Crohn's Disease patients that would benefit from sexual health interventions.

Hypothesis:

Crohn's patients with active perianal fistulas will have decreased sexual drive, performance, and satisfaction than those with Crohn's Disease in remission.

DETAILED DESCRIPTION:
Subject Selection:

Inclusion Criteria Patients in a stable sexual relationship between the ages of 19 and 70 of both sexes with Crohn's disease, as diagnosed based on clinical, radiological, endoscopic or histopathological criteria for a minimum of 6 months will be included in this study. Patients included in this study will have been sexually active in the last 4 weeks.

Exclusion Criteria All patients with known depression will be excluded from the study to prevent confounding the findings.

Patients that qualify for the study will be recruited, and be divided into inactive Crohn's Disease group with no peri-anal fistulas as a control group and an active Crohn's Disease with peri-anal fistula as the study group. Inactive Crohn's Disease patients will be defined as patients with Harvey-Bradshaw scores below 5. Fistula patients will be defined as patients with single or multiple draining fistulas, including perianal fistulas and enterocutaneous fistulas, for at least three months (17).

ELIGIBILITY:
Inclusion Criteria:

* patients in a stable sexual relationship between 19-70 years old with Crohn's Disease
* Crohn's disease diagnosis is based on clinical, radiological, endoscopic or histopathological criteria for a minimum of 6 months
* Patients will have been sexually active in the last 4 weeks.

Exclusion Criteria:

* All patients with known depression will be excluded from the study to prevent confounding the findings.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women ages 19-70 years old with Crohn's disease and sexually active in the last 4 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
CD patients without perianal fistulas will be compared with CD patients with perianal fistulas in terms of the percentage of patients that exhibit our definition of sexual dysfunction. | 1.5 years
  Student t-test will be used to compare the difference between the fistula versus the control group. Statistical analysis will be two tailed and our p value will be set up as p <0.05. We estimate that 30% of patients with CD will have sexual dysfunction, and that 65% of CD patients with peri-anal fistulas will have sexual dysfunction. Therefore, our calculated sample size for both groups will be around 31 patients each for 80% power with an alpha of 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Bressler, MD, Principal Investigator — University of British Columbia
Locations (1):
- Gastroenterology Research Institute, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Thomas E, Koumouvi K, Blotman F. Impotence in a patient with rheumatoid arthritis treated with methotrexate. J Rheumatol. 2000 Jul;27(7):1821-2. No abstract available. PMID 10914881
- [Background] Riba N, Moreno F, Costa J, Olive A. [Appearance of impotence in relation to the use of methotrexate]. Med Clin (Barc). 1996 Apr 13;106(14):558. No abstract available. Spanish. PMID 8656751
- [Background] Ireland A, Jewell DP. Sulfasalazine-induced impotence: a beneficial resolution with olsalazine? J Clin Gastroenterol. 1989 Dec;11(6):711. No abstract available. PMID 2573629
- [Background] Levi AJ, Fisher AM, Hughes L, Hendry WF. Male infertility due to sulphasalazine. Lancet. 1979 Aug 11;2(8137):276-8. doi: 10.1016/s0140-6736(79)90292-7. PMID 88609
- [Background] Sussman A, Leonard JM. Psoriasis, methotrexate, and oligospermia. Arch Dermatol. 1980 Feb;116(2):215-7. PMID 7356357
- [Background] Farouk R, Pemberton JH, Wolff BG, Dozois RR, Browning S, Larson D. Functional outcomes after ileal pouch-anal anastomosis for chronic ulcerative colitis. Ann Surg. 2000 Jun;231(6):919-26. doi: 10.1097/00000658-200006000-00017. PMID 10816636
- [Background] Timmer A, Bauer A, Kemptner D, Furst A, Rogler G. Determinants of male sexual function in inflammatory bowel disease: a survey-based cross-sectional analysis in 280 men. Inflamm Bowel Dis. 2007 Oct;13(10):1236-43. doi: 10.1002/ibd.20182. PMID 17508419
- [Background] El-Tawil AM. Zinc deficiency in men with Crohn's disease may contribute to poor sperm function and male infertility. Andrologia. 2003 Dec;35(6):337-41. doi: 10.1046/j.0303-4569.2003.00588.x. PMID 15018135
- [Background] Timmer A, Bauer A, Dignass A, Rogler G. Sexual function in persons with inflammatory bowel disease: a survey with matched controls. Clin Gastroenterol Hepatol. 2007 Jan;5(1):87-94. doi: 10.1016/j.cgh.2006.10.018. PMID 17234557
- [Background] Moody G, Probert CS, Srivastava EM, Rhodes J, Mayberry JF. Sexual dysfunction amongst women with Crohn's disease: a hidden problem. Digestion. 1992;52(3-4):179-83. doi: 10.1159/000200951. PMID 1459352
- [Background] Timmer A, Kemptner D, Bauer A, Takses A, Ott C, Furst A. Determinants of female sexual function in inflammatory bowel disease: a survey based cross-sectional analysis. BMC Gastroenterol. 2008 Oct 3;8:45. doi: 10.1186/1471-230X-8-45. PMID 18834529
- [Background] Ogilvie JW Jr, Goetz L, Baxter NN, Park J, Minami S, Madoff RD. Female sexual dysfunction after ileal pouch-anal anastomosis. Br J Surg. 2008 Jul;95(7):887-92. doi: 10.1002/bjs.6072. PMID 18551505
- [Background] McKee RF, Keenan RA. Perianal Crohn's disease--is it all bad news? Dis Colon Rectum. 1996 Feb;39(2):136-42. doi: 10.1007/BF02068066. PMID 8620778
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Sands BE, Anderson FH, Bernstein CN, Chey WY, Feagan BG, Fedorak RN, Kamm MA, Korzenik JR, Lashner BA, Onken JE, Rachmilewitz D, Rutgeerts P, Wild G, Wolf DC, Marsters PA, Travers SB, Blank MA, van Deventer SJ. Infliximab maintenance therapy for fistulizing Crohn's disease. N Engl J Med. 2004 Feb 26;350(9):876-85. doi: 10.1056/NEJMoa030815. PMID 14985485
- [Result] Feagins LA, Kane SV. Sexual and reproductive issues for men with inflammatory bowel disease. Am J Gastroenterol. 2009 Mar;104(3):768-73. doi: 10.1038/ajg.2008.90. Epub 2009 Feb 17. PMID 19223893
- [Result] Mekhjian HS, Switz DM, Melnyk CS, Rankin GB, Brooks RK. Clinical features and natural history of Crohn's disease. Gastroenterology. 1979 Oct;77(4 Pt 2):898-906. PMID 381094